CLINICAL TRIAL: NCT04239729
Title: A Randomized Waitlist-controlled Trial of Web-based Acceptance and Commitment Therapy for Hoarding Disorder
Brief Title: Web-based Acceptance and Commitment Therapy for Hoarding Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10223
Record Dates: First submitted 2020-01-13; First posted 2020-01-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Hoarding Disorder
MeSH Terms: conditions — Hoarding Disorder

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned with equal likelihood to receive the website and coaching immediately or to wait for 12 weeks before using the website.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT Website and Coaching Condition (Experimental): Participants will be asked to complete 16 brief self-help website sessions, each taking around 15-20 minutes to finish, twice a week for eight weeks. Website exercises and examples primarily focus on hoarding, although some examples also discuss related mental health concerns such as anxiety, low mood, health behaviors, etc. The sessions use multimedia and are interactive. Participants assigned to the website condition will also receive coaching. The purpose of coaching will be to help participants engage with the website and adhere to the intervention. Coaching will consist of an initial phone call of 10-15 minutes followed by weekly email contact during the 8-week treatment period. Coaches will be graduate students trained in clinical psychology.
  Interventions: Behavioral: ACT Website and Coaching
- Waitlist Condition (No Intervention): Participants assigned to the waitlist will be asked to wait 12 weeks without intervention (access to the website or coaching). They will receive access to the website after 12 weeks, but supportive coaching will not be provided to waitlist participants.

INTERVENTIONS:
Behavioral: ACT Website and Coaching — The ACT website includes sixteen sessions and is designed to teach a series of skills from ACT applied to hoarding. The intervention also includes brief supportive coaching (an initial phone call and weekly support over email).
  Arms: ACT Website and Coaching Condition

SUMMARY:
This study will help to determine if acceptance and commitment therapy delivered as a web-based intervention is a useful treatment for hoarding disorder and evaluate whether or not web-based treatment for hoarding is credible and acceptable. It may also help identify novel processes of change in hoarding treatment such as psychological inflexibility, mindfulness, and self-stigma.

DETAILED DESCRIPTION:
The efficacy of an ACT self-help website for hoarding will be assessed through a randomized, waitlist-controlled trial. Participants will be recruited from within the United States through a variety of channels. Given the need to recruit a targeted sample with clinical levels of hoarding symptoms, online advertisements through Facebook and Google AdWords will be the primary recruitment method. Participants will complete an initial brief screening, provide consent, and then complete a baseline survey. Each of these steps will be completed online and participants will be automatically guided from each step to the next. That is, those who screen as eligible will be automatically directed to an online consent form, and those who provide consent will be automatically directed to begin the initial online baseline survey. They will be randomly assigned automatically upon completing the baseline survey to either use the ACT self-help website and receive supportive coaching for the next 8 weeks, or wait for the next 8 weeks. After 8 weeks, participants will be asked to complete a posttreatment survey. They will be asked to complete a final, follow-up survey after an additional 4 weeks after the posttreatment survey. After the follow-up survey is completed, waitlisted participants will be provided with access to the website. The website will implement a self-help version of ACT. Participants will be asked to complete 16 brief self-help website sessions, each taking around 15-20 minutes to finish, twice a week for eight weeks. Participants assigned to the website condition will also receive coaching.The purpose of coaching will be to help participants engage with the website and adhere to the intervention. Coaching will consist of an initial phone call of 10-15 minutes followed by weekly email contact during the 8-week treatment period. Coaches will be graduate students trained in clinical psychology.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older
2. Living in the USA
3. Seeking help for clutter and/or hoarding
4. Interested in testing a self-help website
5. Scoring at or above the clinical cutoff of 41 on the Saving Inventory-Revised

Exclusion Criteria:

1. 17 years or younger
2. Living outside the USA
3. Not seeking help for clutter and/or hoarding
4. Not interested in testing a self-help website
5. Scoring below 41 on the Saving Inventory-Revised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Saving Inventory-Revised (SI-R; Frost et al., 2004) | Posttreatment (8 weeks after baseline)
  A self-report measure of hoarding symptoms

SECONDARY OUTCOMES:
Sheehan Disability Scale (Sheehan, Harnett-Sheehan, & Raj, 1996) | Posttreatment (8 weeks after baseline) and follow-up (12 weeks after baseline)
  A self-report measure of functional impairment due to symptoms. Higher scores indicate greater impairment. Scores range from 0 to 30.
Clinical Global Impression - Improvement (CGI-I; Guy, 1976). | Posttreatment (8 weeks after baseline) and follow-up (12 weeks after baseline)
  A self-report measure of overall improvement in symptoms
General Health Questionnaire-12 (GHQ-12; Goldberg, 1978) | Posttreatment (8 weeks after baseline) and follow-up (12 weeks after baseline)
  A self-report measure of overall psychological distress
Stigma of hoarding items (Chasson et al., 2018) | Posttreatment (8 weeks after baseline) and follow-up (12 weeks after baseline)
  Seven self-report items assessing stigma towards individuals with hoarding disorder. These items are not a standardized scale but have been used in previous research (Chasson et al., 2018). Three items assess perceived difference (Example: How like or unlike do you think is a person with obsessive-compulsive disorder compared to everyone else in the general population?), three items assess disdain (Example: How good or bad do you think is a person with hoarding disorder compared to everyone else in the general population?) and one item assesses blame: How responsible do you think a person with serious mental illness is for his or her condition?
Acceptance and Action Questionnaire for Hoarding (AAQH; Krafft et al., in press) | Posttreatment (8 weeks after baseline) and follow-up (12 weeks after baseline)
  A self-report measure of hoarding-related psychological inflexibility
Five-Facet Mindfulness Questionnaire - Acting with Awareness (FFMQ-AA; Baer, Smith, Hopkins, Krietemeyer, & Toney, 2006) | Posttreatment (8 weeks after baseline) and follow-up (12 weeks after baseline)
  A self-report measure of the acting with awareness facet of mindfulness
Valuing Questionnaire-Progress (VQ-Progress; Smout, Davies, Burns, & Christie, 2014) | Posttreatment (8 weeks after baseline) and follow-up (12 weeks after baseline)
  A self-report measure of progress toward personal values
Credibility/Expectancy Questionnaire (CEQ; Devilly & Borkovec, 2000). | After using first website session (approximately 0-1 weeks after baseline)
  A self-report measure of the perceived credibility of and expectations toward a treatment. Only administered to treatment condition
System Usability Scale (Tullis & Albert, 2008) | Posttreatment (8 weeks after baseline)
  A self-report measure of usability of a technological system. Only administered to treatment condition. High scores indicated greater usability, and scores range from 0 to 100.
Treatment Evaluation Inventory-Short Form (TEI-SF; Kelley, Heffer, Gresham, & Elliott, 1989). | Posttreatment (8 weeks after baseline)
  A self-report measure of treatment acceptability. Only administered to treatment condition
Novel satisfaction item 1 | Posttreatment (8 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "Overall, I was satisfied with the quality of the program." This is a novel satisfaction item specific to this study. Only administered to treatment condition
Novel satisfaction item 2 | Posttreatment (8 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "The program was helpful to me." This is a novel satisfaction item specific to this study. Only administered to treatment condition
Novel satisfaction item 3 | Posttreatment (8 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "The program was easy to use." This is a novel satisfaction item specific to this study. Only administered to treatment condition
Novel satisfaction item 4 | Posttreatment (8 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "I felt the program was made for someone like me." This is a novel satisfaction item specific to this study. Only administered to treatment condition
Novel satisfaction item 5 | Posttreatment (8 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "I would recommend the program to other people with a clutter and/or hoarding problem." This is a novel satisfaction item specific to this study. Only administered to treatment condition
Novel satisfaction item 6 | Posttreatment (8 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "The psychological skills taught (ex. mindfulness, opening up) were helpful to me." This is a novel satisfaction item specific to this study. Only administered to treatment condition
Novel satisfaction item 7 | Posttreatment (8 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "The practice exercises (ex. discarding, goal setting) were helpful to me." This is a novel satisfaction item specific to this study. Only administered to treatment condition
Novel satisfaction item 8 | Posttreatment (8 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "This treatment fit well with my goals." This is a novel satisfaction item specific to this study. Only administered to treatment condition
Novel satisfaction item 9 | Posttreatment (8 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "Overall, I was satisfied with the coaching that I received." This is a novel satisfaction item specific to this study. Only administered to treatment condition
Novel satisfaction item 10 | Posttreatment (8 weeks after baseline)
  Participants will be asked to rate agreement from 1 (Strongly disagree) to 6 (Strongly agree) with the statement "The website would have been just as useful without a coach." This is a novel satisfaction item specific to this study. Only administered to treatment condition
Novel satisfaction item 11 | Posttreatment (8 weeks after baseline)
  Participants will be asked an open-ended question to gather qualitative feedback on the intervention. Only assigned to treatment condition. The question is, "What did you like best about the Making Space program?"
Novel satisfaction item 12 | Posttreatment (8 weeks after baseline)
  Participants will be asked an open-ended question to gather qualitative feedback on the intervention. Only assigned to treatment condition. The question is, "What was the most important thing you learned from the Making Space program?"
Novel satisfaction item 13 | Posttreatment (8 weeks after baseline)
  Participants will be asked an open-ended question to gather qualitative feedback on the intervention. Only assigned to treatment condition. The question is, "What did you like least about the Making Space Program? Why did you like this the least?"
Novel satisfaction item 14 | Posttreatment (8 weeks after baseline)
  Participants will be asked an open-ended question to gather qualitative feedback on the intervention. Only assigned to treatment condition. The question is, "Do you have any other comments or suggestions regarding our Making Space program?"

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Levin, PhD, Principal Investigator — Utah State University
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Frost RO, Steketee G, Grisham J. Measurement of compulsive hoarding: saving inventory-revised. Behav Res Ther. 2004 Oct;42(10):1163-82. doi: 10.1016/j.brat.2003.07.006. PMID 15350856
- [Background] Sheehan DV, Harnett-Sheehan K, Raj BA. The measurement of disability. Int Clin Psychopharmacol. 1996 Jun;11 Suppl 3:89-95. doi: 10.1097/00004850-199606003-00015. PMID 8923116
- [Background] Guy, W. (1976). Clinical Global Impressions ECDEU Assessment Manual for Psychopharmacology, Revised (DHEW Publ. No. ADM 76-338). Rockville, MD: National Institute of Mental Health.
- [Background] Goldberg, D. (1978). Manual of the GHQ. Windsor: NFER.
- [Background] Chasson, G. S., Guy, A. A., Bates, S., & Corrigan, P. W. (2018). They aren't like me, they are bad, and they are to blame: A theoretically-informed study of stigma of hoarding disorder and obsessive-compulsive disorder. Journal of Obsessive-Compulsive and Related Disorders, 16, 56-65. http://doi.org/10.1016/j.jocrd.2017.12.006
- [Background] Krafft, J., Ong, C. W., Twohig, M. P., & Levin, M. E. (In press). Assessing psychological inflexibility in hoarding: The Acceptance and Action Questionnaire for Hoarding (AAQH). Journal of Contextual Behavioral Science.http://doi.org/10.1016/j.jcbs.2018.08.003
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Smout, M., Davies, M., Burns, N., & Christie, A. (2014). Development of the Valuing Questionnaire (VQ). Journal of Contextual Behavioral Science, 3, 164-172. http://doi.org/10.1016/j.jcbs.2014.06.001
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Tullis, T., & Albert, W. (2008). Measuring the user experience. San Francisco, CA: Morgan Kaufmann.
- [Background] Kelley, M. L., Heffer, R. W., Gresham, F. M., & Elliott, S. N. (1989). Development of a modified treatment evaluation inventory. Journal of Psychopathology and Behavioral Assessment, 11, 235-247.